CLINICAL TRIAL: NCT06024174
Title: Phase 1/2 Open-label Study of BMS-986466 in Combination With Adagrasib With or Without Cetuximab in Participants With KRAS G12C-mutant Advanced Solid Tumors
Brief Title: A Study of BMS-986466 With Adagrasib With or Without Cetuximab in Participants With Kirsten Rat Sarcoma Virus Glycine 12 to Cysteine (KRAS G12C)-Mutant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA126-0015; 2023-505070-15 (EudraCT Number)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: BMS-986466; KRAS G12C-mutant; Pancreatic duct adenocarcinoma; Biliary tract cancer; Colorectal cancer; Non-small cell lung cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — adagrasib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: DDI Cohort (Experimental)
  Interventions: Drug: BMS-986466; Drug: Adagrasib
- Part 1: Dose Escalation (Experimental)
  Interventions: Drug: BMS-986466; Drug: Adagrasib; Drug: Cetuximab
- Part 2: Dose Expansion (Experimental)
  Interventions: Drug: BMS-986466; Drug: Adagrasib; Drug: Cetuximab

INTERVENTIONS:
Drug: BMS-986466 — Specified dose on specified days
  Other Names: BBP-398; IACS-15509
Drug: Adagrasib — Specified dose on specified days
  Other Names: MRTX849; KRAZATI®
Drug: Cetuximab — Specified dose on specified days
  Other Names: Erbitux®
  Arms: Part 1: Dose Escalation; Part 2: Dose Expansion

SUMMARY:
The purpose of this study is to find a safe, tolerable, and efficacious dose of BMS-986466 when given orally, in combination with adagrasib with or without cetuximab in participants with advanced KRAS G12C-mutant non-small cell lung cancer (NSCLC), pancreatic duct adenocarcinoma (PDAC), biliary tract cancer (BTC), or colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

Part 1:

* Individuals with a confirmed diagnosis of advanced KRAS G12C mutant NSCLC, CRC, PDAC and BTC that has spread to other parts of the body and cannot be removed surgically, may or may not have received previous treatment with KRAS G12C inhibitors.
* For NSCLC and CRC: Individuals must have a documented KRAS G12C mutation status from NYS or FDA approved/cleared or CE marked test or, when such result is not available, positive KRAS G12C mutation status should be confirmed by a central laboratory in blood sample collected at the time of screening.
* For PDAC and BTC: Participants must have a documented KRAS G12Cmutation from NYS or FDA-approved/cleared, or CE-marked test and blood samples will be collected only for retrospective testing.
* Are relapsed or refractory to available standard of care treatments.

Part 2:

* Individuals with a confirmed diagnosis of advanced KRAS G12C-mutant NSCLC (Part 2A) or CRC (Part 2B) that has spread to other parts of the body and cannot be removed surgically and have not received previous treatment with KRAS inhibitors.
* Individuals must have a documented KRAS G12C mutation from FDA or NYS approved/ cleared or CE marked test or, when such result is not available, positive KRAS G12C mutation status should be confirmed by a central laboratory in blood sample and /or tumor samples collected at the time of screening or from archival biopsies (less than 1 year old).
* Have failed or disease recurrence or are not able to tolerate after at least 1 pervious line of therapy.

Key Exclusion Criteria:

* Have tumors with known BARF V600X, PTPN11 or KRASQ61X mutations.
* Have or any significant heart disease or condition.
* Receiving any medications that are substrate of CYP3A4 or inducers and/ or inhibitors

Note: Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (4):
  - Local Institution - 0047, Los Angeles, California
  - Local Institution - 0040, Athens, Georgia
  - Local Institution - 0025, Hackensack, New Jersey
  - Local Institution - 0008, Morristown, New Jersey
- Local Institution - 0053, Westmead, New South Wales, Australia
- Local Institution - 0083, Helsinki, Finland
- Local Institution - 0020, Lille, France
- Israel (2):
  - Local Institution - 0082, Petah Tikva, Central District
  - Local Institution - 0081, Tel Aviv, Tell Abīb

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was early terminated and participants were not enrolled in Part 1A and 1B (Dose Escalation) and Part 2A and 2B (Dose Expansion).
Groups:
- Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID: Participants with KRAS G12C-mutant Advanced Solid Tumors were treated with a single dose of BMS-986466 10 mg orally (PO) on Cycle 1 Day 1 and Day 9 and followed by regular administration from Cycle 3 Day 1 till study discontinuation. Participants were also administered with adagrasib 400 mg twice a day (BID) starting on Cycle 1 Day 4.
Period: Overall Study
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Started | 5
Completed | 0
Not Completed | 5
Not completed — Other Reasons | 1
Not completed — Study terminated by Sponsor | 4

BASELINE CHARACTERISTICS:
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 1
  WHITE | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicity (DLTs)
Description: A DLT was defined as:
  * Death not related to disease progression
  * Grade (Gr) 4 (Life-threatening) neurotoxicity
  * Gr 3 (Severe) neurotoxicity of greater than 7 days
  * Gr 3 neurotoxicity does not revert to baseline within 28 days of the start date of the Grade 3 event
  * Seizures of grade that do not resolve within 7 days
  * Gr 4 cytokine release syndrome (CRS) that does not resolve to less than or equal to Gr 3 within 3 days
  * Gr 3 CRS that does not resolve to less than or equal to Grade 2 within 7 days
  * Any increase in aspartate aminotransferase (AST) or ALT > 3 Ã- ULN and concurrent increase in total bilirubin > 2 Ã- ULN that is unrelated to CRS and has no other probable reason to explain the combination of increases
  * Any other Gr 3 or 4 event deemed unexpected by the Investigator and considered a DLT upon evaluation by the safety review committee
Time Frame: Cycle 1 (Each cycle consist of 28 days)
Population: All treated participants were considered DLT evaluable if they complete ≥ 75% of all planned doses of BMS-986466 and adagrasib without experiencing a DLT or experience a DLT after receiving at least 1 dose of BMS-986466 and adagrasib. Participants were not enrolled in Part 1a, 1b. Prespecified to be collected for Part 1 only
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: All treated population include all participants who received at least 1 dose of study intervention. Participants were not enrolled in Part 1a, 1b. Prespecified to be collected for Part 1 only
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
Participants | 4

3. Primary Outcome: Part 1: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability or permanent damage, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: From first dose until 30 days after last dose (Up to approximately 3 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
Participants | 1

4. Primary Outcome: Part 1: Number of Participants With AEs Leading to Discontinuation
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatmen
Time Frame: From first dose until 30 days after last dose (Up to approximately 3 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
Participants | 0

5. Primary Outcome: Part 1: Number of Participants Who Died
Description: Death due to any cause was assessed.
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
Participants | 0

6. Primary Outcome: Part 2 Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Objective Response Rate (ORR) is defined as the percentage of participants with a confirmed Best overall response of Complete Response (CR) or Partial Response (PR) by RECIST v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 5 months)
Population: All treated population include all participants who received at least 1 dose of study intervention. Participants were not enrolled in Part 2, hence participants analyzed is 0. Prespecified to be collected for Part 2 only
Groups:
- Part 2A: Part 2A were planned to evaluate BMS-986466 in combination with adagrasib in KRAS G12C-mutant (G12C inhibitor treatment-naïve) NSCLC participants.
- Part 2B: Part 2B were planned to evaluate BMS-986466 in combination with adagrasib with or without cetuximab in KRAS G12C-mutant(G12C inhibitor treatment-naïve) CRC participants.
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax)
Description: Blood samples were collected to assess adequate PK profiles. Participants were not enrolled in Part 1a, 1b.
Time Frame: Cycle 1 Day 1 (Each cycle consist of 28 days)
Population: Pharmacokinetic (PK) evaluable population is a subset of PK participants (all participants who received at least 1 dose of BMS-986466 and/or adagrasib and had any available concentration-time data) which consist of all participants in the PK population with adequate PK profiles. Prespecified to be collected for Part 1 only
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
ng/mL | NA (NA) — No participants had adequate PK profiles (below lower limit of quantification).

8. Secondary Outcome: Part 1: Time to Maximum Concentration (Tmax)
Description: Blood samples were collected to assess adequate PK profiles. Participants were not enrolled in Part 1a, 1b.
Time Frame: Cycle 1 Day 1 (Each cycle consist of 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
hours | NA (NA) — No participants had adequate PK profiles (below lower limit of quantification).

9. Secondary Outcome: Part 1: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-T])
Description: Blood samples were collected to assess adequate PK profiles. Participants were not enrolled in Part 1a, 1b.
Time Frame: Cycle 1 Day 1 (Each cycle consist of 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
Number analyzed (Participants) | 5
mcg*hr/mL | NA (NA) — No participants had adequate PK profiles (below lower limit of quantification).

10. Secondary Outcome: Part 2-Progression-free Survival (PFS) Assessed by BICR as Per RECIST v1.1
Description: Progression-Free Survival then (PFS) is defined as the time between the date of randomization and the date of first documented disease progression, based on Investigator assessments (per RECIST v1.1), or death due to any cause, whichever occurs first Calculated using Kaplan-Meier estimates. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 5 months)
Population: Participants were not enrolled in Part 2 arm, hence participants analyzed is 0. Prespecified to be collected for Part 2 only
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Part 2- Disease Control Rate (DCR) Assessed by BICR as Per RECIST v1.1
Description: Disease Control Rate (DCR) (as per Recists v1.1) is defined as the number of randomized participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD), based on BICR assessments divided by the number of all randomized participants.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Part 2- Duration of Response (DOR) Assessed by BICR as Per RECIST v1.1
Description: Duration of objective response (DoR) is defined as the time between the date of first confirmed response (CR or PR) to the date of the first documented tumor progression (per RECIST 1.1) per BICR assessment, or death due to any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part 2- Time to Response (TTR)
Description: Time to response (TTR) is defined as the time, in months, from randomization to the first objective documentation of PR or better assessed per BICR.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
Time Frame: From randomization untill disease progression or death, whichever occurs first (up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part 2- Number of Participants With Adverse Events (AEs)
Description: as for outcome 2
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part 2- Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability or permanent damage, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 2- Number of Participants With AEs Leading to Discontinuation
Description: as for outcome 2
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part 2- Number of Participants Who Died
Description: Death due to any cause was assessed.
Time Frame: From first dose until 100 days after last dose (Up to approximately 5 months)
Population: as for outcome 10
Arm/Group | Part 2A | Part 2B
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part 1a and 1b - Changes From Baseline in Pharmacodynamic Biomarker
Description: Blood samples were collected for assessing pharmacodynamic parameters.
Time Frame: Baseline and Cycle 1 Day 1 (Each cycle consist of 28 days)
Population: All treated participants with available biomarker data. Participants were not enrolled in Part 1a and 1b arm, hence participants analyzed is 0. Prespecified to be collected for Part 1A and 1B only.
Groups:
- Part 1A: Part 1A consist of dose escalation of BMS-986466 in combination with adagrasib in KRAS G12C-mutant NSCLC, PDAC, BTC, and CRC.
- Part 1B: Part 1B was planned to evaluate the dose escalation of BMS-986466 in combination with adagrasib plus Cetuximab in KRAS G12C-mutant CRC.
Arm/Group | Part 1A | Part 1B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, and serious and non-serious adverse events were collected from from first dose until 100 days after last dose (Up to approximately 5 months).
Description: All treated population include all participants who received at least 1 dose of study intervention.
Arm/Group | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID (N=5)
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Drug-Drug Interaction (DDI) - BMS986466 10 MG + Adagrasib 400MG BID (N=5)
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Somnolence (Nervous system disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT06024174/Prot_SAP_000.pdf